CLINICAL TRIAL: NCT01892540
Title: Positron Mammographic Imaging (PMI)
Brief Title: PET/CT or PET/MRI in Measuring Tumors in Patients Undergoing Clinical Imaging or With Newly Diagnosed Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE15112; NCI-2013-00938 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PMI TECH 12-050 (Other: University Hospitals)
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Breast Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1: Standard positioning device (Experimental): Patients undergo clinical FDG-PET/CT followed by prone breast PET/CT and/or prone breast PET/MRI with or without DTPA.
  Interventions: Diagnostic Test: positron emission tomography/computed tomography; Diagnostic Test: PET/MRI
- Cohort 2: New positioning device (Experimental)
  Interventions: Diagnostic Test: positron emission tomography/computed tomography; Diagnostic Test: PET/MRI; Device: Position Device
- Cohort 3: Current positioning device until new is available (Experimental)
  Interventions: Diagnostic Test: positron emission tomography/computed tomography; Diagnostic Test: PET/MRI; Device: Position Device

INTERVENTIONS:
Diagnostic Test: positron emission tomography/computed tomography — Undergo PET/CT
Diagnostic Test: PET/MRI — Undergo PET/MRI positron emission tomography/magnetic resonance imaging hybrid imaging
Device: Position Device
  Arms: Cohort 2: New positioning device; Cohort 3: Current positioning device until new is available

SUMMARY:
This clinical trial studies positron emission tomography (PET)/computed tomography (CT) or PET/magnetic resonance imaging (MRI) in measuring tumors in patients undergoing clinical imaging or with newly diagnosed breast cancer. New diagnostic procedures, such as PET/CT or PET/MRI, may be more effective than MRI alone in measuring tumors in patients undergoing clinical imaging or with newly diagnosed breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To improve visualization of tumors by developing better image reconstruction and correction methods.

II. To revise the positioning devices and, if necessary, scanner table to fit a wider size range of women.

OUTLINE:

Patients undergo clinical fludeoxyglucose F-18 (FDG)-PET/CT followed by prone breast PET/CT and/or prone breast PET/MRI with or without gadopentetate dimeglumine (DTPA).

ELIGIBILITY:
Inclusion Criteria:

* [Cohorts 1 and 2] Female patients who are referred by their physician to have a clinical PET/CT
* [Cohort 3] Patients referred for clinical breast dynamic contrast-enhanced (DCE)-MRI for recently diagnosed breast cancer
* Normal kidney function for subjects that will receive magnetic resonance (MR) contrast agent as part of their clinical imaging
* For subjects for whom MR contrast agent is to be administered, University Hospitals (UH) policy 8.17.26 will be applied

  * The following guidelines will be followed when a patient or patient representative responds "yes" to questions on the MRI history sheet 'Are you on dialysis, history of kidney failure, end stage renal disease, chronic liver disease, or are you a peri-liver transplant patient':

    * The patient must have a serum creatinine value available within three (3) weeks prior to the injection of gadolinium
    * Calculate an estimated glomerular filtration rate (eGFR) based on serum creatinine; if the eGFR is less than 30 the attending radiologist must discuss the risks and benefits of administering gadolinium with the referring physician and patient; the collective judgment of the patient, radiologist and referring physician must be in agreement to proceed with the injection of gadolinium
    * Calculated eGFR in range of 31-59 requires the judgment of the attending radiologist whether to discuss gadolinium administration with referring physician and patient or whether to directly use or hold the contrast agent
    * If an eGFR is greater than 60, gadolinium may be administered without further physician or patient discussion
    * Gadolinium administration is limited to single dose at 0.1mmol/kg; Omniscan should not be used
    * Technologist will document radiologist decision to administer gadolinium on the MRI history sheet; radiologist will document decision and consultation with the referring physician and patient in the MRI report
    * PERITONEAL DIALYSIS PATIENTS:

      * No gadolinium will be administered unless the patient has been scheduled for hemodialysis within 24 hours following the injection of gadolinium; technologist will determine eGFR and follow above guidelines; dialysis will be scheduled by the referring physician
    * HEMODIALYSIS PATIENTS:

      * No gadolinium will be administered unless the patient has been scheduled for hemodialysis within 24 hours following the injection of gadolinium; no determination of eGFR is necessary; radiologist will assume eGFR less than 30 and follow above guidelines; dialysis will be scheduled by the referring physician
* Ability to provide informed consent

Exclusion Criteria:

* Subjects who do not meet all of the above inclusion criteria
* Subjects unwilling or unable to sign the informed consent form
* Subjects who are cognitively impaired and thus unable to give informed consent
* Subjects unable to undergo MR scanning due to exclusion via University Hospitals Case Medical Center (UHCMC) MR restrictions (e.g. certain implanted metallic or electronic devices)
* Subjects who are pregnant
* Subjects that are too large to fit comfortably into the PET/MR on the breast coil; for cohort 1 only we will accept a maximum of 10 subjects that are too large for the PET/MRI to acquire a prone PET/CT but without the paired PET/MR

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Plecha, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2: New Positioning Device; Cohort 3: Current Positioning Device Until New is Available: positron emission tomography/computed tomography: Undergo PET/CT
  PET/MRI: Undergo PET/MRI positron emission tomography/magnetic resonance imaging hybrid imaging
  Position Device
Period: Overall Study
Arm/Group | Cohort 1: Standard Positioning Device | Cohort 2: New Positioning Device | Cohort 3: Current Positioning Device Until New is Available
Started | 15 | 0 | 28
Completed | 15 | 0 | 25
Not Completed | 0 | 0 | 3
Not completed — Did not complete PET/MRI | 0 | 0 | 2
Not completed — Did not fit in scanner | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: No participants accrued to cohort 2
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Standard Positioning Device | Cohort 2: New Positioning Device | Cohort 3: Current Positioning Device Until New is Available | Total
Number analyzed (Participants) | 15 | 0 | 28 | 43
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 3 | 0 | 4 | 7
  40-49 years | 3 | 0 | 5 | 8
  50-59 years | 2 | 0 | 10 | 12
  60-69 years | 4 | 0 | 7 | 11
  70-79 years | 3 | 0 | 2 | 5
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 11 | 0 | 26 | 37
  Gender: Unknown | 4 | 0 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 14 | 0 | 25 | 39
  Unknown or Not Reported | 1 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 7 | 8
  White | 12 | 0 | 19 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 |  | 28 | 43

OUTCOME MEASURES:

1. Primary Outcome: Attenuation Correction for PET/MRI, Assessed Using Standard Uptake Values (SUVs) (Cohorts I & II)
Description: Uptake and attenuation correction of PET/MRI and PET/CT will be examined by comparing SUVs of the two methods. The proportions of subjects with SUV of the PET/MR within 5%, 10%, and 20% of the SUV from PET/CT will be estimated with exact 95% confidence intervals.
Time Frame: 1 yr from study start
Population: No data available - SUV data do not exist for Cohort I and cohort II was never conducted.
Arm/Group | Cohort 1: Standard Positioning Device | Cohort 2: New Positioning Device | Cohort 3: Current Positioning Device Until New is Available
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Attenuation Correction for PET/CT, Assessed Using SUVs (Cohorts I & II)
Description: as for outcome 1
Time Frame: 1 yr from study start
Population: No data available - SUV data do not exist for Cohort I and cohort II was never conducted.
Arm/Group | Cohort 1: Standard Positioning Device | Cohort 2: New Positioning Device | Cohort 3: Current Positioning Device Until New is Available
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Comparison of Specificity Rates of Fused FDG-PET/MRI (Cohort III)
Description: McNemar's test or a generalized estimating equations logistic regression model with patient as the cluster used to compare specificity rates of the new technology versus current technology (MRI alone), restricting analysis to true negative lesions. Utilizing 3 different combinations of scan parameters to determine which combination has the highest specificity. Single parameter: DCE-MRI is the gold standard to which the two parameter and three parameter rows are compared.
  Combinations include:
  Single parameter: DCE-MRI Two Parameter A: DCE-MRI and DWI ADC Two Parameter B: DCE-MRI and FDG-PET Three Parameter: DCE-MRI, DWI ADC, FDG-PET
Time Frame: 1 yr from study start
Population: Participants in cohort 3 that completed scans.
Measure: Mean (Full Range); unit: percent of specificity
Arm/Group | Cohort 1: Standard Positioning Device | Cohort 2: New Positioning Device | Cohort 3: Current Positioning Device Until New is Available
Number analyzed (Participants) | 0 | 0 | 25
percent of specificity
  Single parameter: DCE-MRI |  |  | 0 [0 to 0]
  Two Parameter A: DCE-MRI and DWI ADC |  |  | 89 [52 to 100]
  Two Parameter B: DCE-MRI and FDG-PET |  |  | 89 [52 to 100]
  Three Parameter: DCE-MRI, DWI ADC, FDG-PET |  |  | 100 [66 to 100]

4. Primary Outcome: Sensitivity of PET/CT and PET/MRI (Cohort III)
Description: McNemar's test or a generalized estimating equations logistic regression model with patient as the cluster used to compare sensitivity rates of the new technology versus current technology (MRI alone), restricting analysis to true negative lesions. Utilizing 3 different combinations of scan parameters to determine which combination has the highest sensitivity.
  Combinations include:
  Single parameter: DCE-MRI Two Parameter A: DCE-MRI and DWI ADC Two Parameter B: DCE-MRI and FDG-PET Three Parameter: DCE-MRI, DWI ADC, FDG-PET
Time Frame: 1 yr from study start
Population: Participants in cohort 3 that completed scans.
Measure: Mean (Full Range); unit: percent sensitivity
Arm/Group | Cohort 1: Standard Positioning Device | Cohort 2: New Positioning Device | Cohort 3: Current Positioning Device Until New is Available
Number analyzed (Participants) | 0 | 0 | 25
percent sensitivity
  Single parameter: DCE-MRI |  |  | 100 [100 to 100]
  Two Parameter A: DCE-MRI and DWI ADC |  |  | 95 [83 to 100]
  Two Parameter B: DCE-MRI and FDG-PET |  |  | 86 [71 to 100]
  Three Parameter: DCE-MRI, DWI ADC, FDG-PET |  |  | 85 [70 to 94]

ADVERSE EVENTS:
Time Frame: Adverse vents and other safety parameters monitored throughout study for up to 1 yr from study start
Description: No participants were enrolled in cohort 2, so no participants are at risk for adverse vents.
Arm/Group | Cohort 1: Standard Positioning Device | Cohort 2: New Positioning Device | Cohort 3: Current Positioning Device Until New is Available
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/0 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/0 | 0/28
Other Adverse Events (participants affected / at risk) | 0/15 | 0/0 | 0/28

LIMITATIONS AND CAVEATS:
Cohort 1 was not completed (15 of 40 participants) and cohort 2 was not collected because of recruitment issues.

Imaging data was collected for available participants but SUV data were not collected from images due to low recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes